CLINICAL TRIAL: NCT02372812
Title: Analgesic Effects Of Dexamethasone; Its Use To Reduce Post Operative Pain Scores: A Double Blinded Randomised Controlled Clinical Trial
Brief Title: Analgesic Effects Of Dexamethasone; Its Use To Reduce Post Operative Pain Scores
Acronym: DOPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Medical doctor, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 206000541
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Pain
Keywords: effect of dexamethasone; general surgery; post operative
MeSH Terms: conditions — Pain | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group1 (Active Comparator): 12 mg( 3 mls) of dexamethasone given 15 mins after induction of anesthesia
  Interventions: Drug: dexamethasone
- group2 (Placebo Comparator): 3 mls of placebo( normal saline) given 15 mins after induction of anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dexamethasone — 12 mg of dexamethasone
  Arms: group1
Drug: Placebo
  Arms: group2

SUMMARY:
A randomised controlled clinical trial to assess the effect of intraoperative dexamethasone on the 24 hour post operative pain scores of adult patients in Mulago hospital undergoing mastectomies, laparotomies and thyroidectomies. The adverse effects of dexamethasone at this dose were also assessed for.

DETAILED DESCRIPTION:
RESEARCH QUESTION TO BE ADDRESSED BY THIS RESEARCH Does intraoperative dexamethasone 12mg reduce 24 hour post-operative pain scores of adult patients undergoing elective laparotomies, thyroidectomies and mastectomies in Mulago hospital RATIONALE FOR THE RESEARCH The treatment of acute post-operative pain is an important health care issue. Inspite of that, its under treatment has been widely recognised over the past two decades. A variety of cultural, attitudinal, religious, educational, political and logistical reasons can be attributed to this and there are a variety of physiological and psychological side effects of this pain.

Dexamethasone is a cheap and readily available drug in Uganda and it has been shown to have analgesic properties.

However, only a few studies have been done to assess these analgesic effects and they have majorly been in tonsillectomies and cardiac surgery. A few such studies have been done on general surgery patients. Most of these studies have been done outside Africa and yet they have demonstrated positive results with regards to optimising analgesia and reducing the post-operative opioid requirements of patients.

This study is yet to be done in Uganda and all the available literature may not necessarily apply to this setting.

GENERAL OBJECTIVE To study the effect of intraoperative dexamethasone 12 mg versus placebo on 24 hour post-operative pain scores of adult patients undergoing elective laparotomies, mastectomies and thyroidectomies in Mulago hospital.

SPECIFIC OBJECTIVES PRIMARY OBJECTIVE To compare the 24 hour post-operative pain scores after intraoperative dexamethasone 12mg versus placebo in adult patients undergoing elective laparotomies, mastectomies and thyroidectomies in Mulago hospital.

SECONDARY OBJECTIVE To compare the adverse events associated with intraoperative dexamethasone 12mg versus placebo in adult patients undergoing elective laparotomies, mastectomies and thyroidectomies in Mulago hospital.

METHODS Study design: a phase 2 prospective randomized, double blinded, placebo-controlled trial Study site: Mulago National Refferal Hospital. Study population: Adult patients undergoing elective laparotomies, mastectomies and thyroidectomies in Mulago hospital, who meet the inclusion criteria and consent to participate in the study.

Inclusion criteria: Patients scheduled for mastectomies, laparotomies and thyroidectomies that have given informed consent to participate, ASA I & II, patients that have none or have mild to moderate systemic illness, Adult patients, above 18 years old.

Exclusion criteria: Patients with Cushing's disease or Cushing's syndrome, Patients with diabetes mellitus, Systemic infection, Previous history of TB infection.

Randomization: block randomization Blinding: double blinded Sample size: 170 patients

Study procedure:

1. Premedication consisted of midazolam and fentanyl .
2. Anaesthesia was induced using intravenous propofol or thiopental.
3. Maintenance of anaesthesia was done using inhalation anaesthesia i.e isoflurane or sevoflurane.
4. The intervention (dexamethasone or placebo) was given 15 minutes following induction of anaesthesia.
5. 30 minutes prior to the end of the procedure, an opioid (morphine) was given intravenously for post operative pain management in the immediate post operative period.
6. Post-operative pain was managed using tramadol or pethidine.
7. Breakthrough pain was managed using intravenous diclofenac as the drug of choice or intravenous paracetamol for those who cannot tolerate opioids.
8. The patients' pain scores were assessed in the post anaesthesia care unit before being discharged to their parent wards.
9. A research assistant was allocated to these patients while on the ward, to ensure timely administration of analgesia as well as the management of breakthrough pain.
10. The pain scores were assessed at 12 and 24 hours, by research assistants who will have been trained on how to administer the numerical rating scale. Their pain scores were assessed using this tool and the adverse reactions assessed.

RISKS OR BENEFITS TO SUBJECTS This is a minimal risk study. There have been no demonstrated risks of the drug at these doses. All patients who might react to the drug will be eliminated from the study.

COMPENSATION/REIMBURSEMENT No patient was expected to pay for this study. Patients were not reimbursed for participating in the study.

CONSENT informed consent was sought from the patients prior to surgery. CONFIDENTIALITY ASSURANCES Patient names and in patient numbers were not collected in order to ensure utmost confidentiality. The other data that was collected was safely stored on multiple soft copies and storage devices in separate places, as were the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* • Patients scheduled for mastectomies, laparotomies and thyroidectomies that have given informed consent to participate.

  * ASA I & II, patients that have none or have mild to moderate systemic illness.
  * Adult patients, above 18 years old.

Exclusion Criteria:

* • Patients with Cushing's disease or Cushing's syndrome

  * Patients with diabetes mellitus
  * Systemic infection
  * Previous history of TB infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Post- operative pain scores of the patients using the numerical rating scale, that grades pain from 1-10. The patients will have this scale explained to them. This will be done 24 hours following administration of intraoperative dexamethasone. | 1 year
  pain scores assessed using the numerical rating scale, at three points i.e the PACU, 12 and 24 hours post operatively

SECONDARY OUTCOMES:
: Adverse effects of the dexamethasone | 1 year
  patients were asked if they had got any drug reactions, their temperatures and glucose levels were assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Mulago Hospital National Refferal, surgical wards, Kampala, Uganda